CLINICAL TRIAL: NCT00863226
Title: A Randomized, Double-Blind, Sham-Stimulation Controlled Study of the Application of Magnetic Fields Using the Resonator Device for the Treatment of Parkinson's Disease: Phase Three Clinical Trial Protocol
Brief Title: Study of the Application of Magnetic Fields for the Treatment of Parkinson's Disease
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: pico-tesla Magnetic Therapies, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 09026-01
Record Dates: First submitted 2009-03-13; First posted 2009-03-17 (Estimated); Last update posted 2011-12-14 (Estimated); Status verified 2011-12

CONDITIONS: Parkinson's Disease; Quality of Life
Keywords: Quality of Life issues in Parkinson's disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

INTERVENTIONS:
Device: Resonator Device — Application of Magnetic Fields Using the Resonator Device

SUMMARY:
The purpose of this study is to see if a device called the Resonator can help to improve aspects of health and quality of life that are relevant to patients with Parkinson's disease.

DETAILED DESCRIPTION:
This clinical trial will evaluate a new non-invasive, non-significant risk, device therapy as an adjuvant symptomatic treatment for some of the signs and or symptoms of Parkinson's Disease (PD). The device utilizes patented technology involving extremely low level electromagnetic fields.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic Parkinson's Disease
* Stable optimized anti-PD drugs for at least 4 weeks
* PDQ-39 Summary Index between 15 and 45
* Ambulatory
* Willing to maintain regular medication regime throughout study
* Able to abstain from starting in new treatments to improve PD symptoms during course of study.
* No prior surgical interventions for Parkinson's Disease
* Non-demented
* Minimum of 30 years of age, but not older than 85
* Capable of giving full written consent

Exclusion Criteria:

* Atypical Parkinsonism such as progressive supranuclear palsy, multiple system atrophy, CBDG etc.
* Subjects may not have any of the following: active brain tumor, strokes, hydrocephalus, any other neurologic or non-neuro problem which may affect symptomatic expression of patients parkinsonism.
* Consumption of medications that can produce drug induced parkinsonism
* Chronic pain not associated with PD
* Current or past history of major psychiatric disturbance
* No typical or non-typical anti-psychotics for treatment of drug induced psychosis.
* Chronic fatigue
* Epilepsy or history of epilepsy
* Seizures or taking medication for epilepsy
* HIV or other autoimmune disorders
* History of ECT
* Uncontrolled hypertension
* Advanced pulmonary disease
* Unstable cardiac disease
* Prior surgical interventions for Parkinson's disease
* Prosthetics or implants comprised of ferrous metals
* Pacemaker, vagus nerve stimulators, or other functional electrical stimulators such as those commonly used for pain
* Pregnant, breast feeding or planning pregnancy prior to study end
* Dementia, developmental disability, psychiatric disorder or other cognitive impairment
* Any significant medical condition that may require alteration of medical therapy during the study, or major medical condition which may interfere with the study activity.

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2009-03; Primary Completion 2012-01 (Estimated); Study Completion 2012-01 (Estimated)

PRIMARY OUTCOMES:
Change in PDQ-39 single index score | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Rajeev Kumar, MD, Principal Investigator; Jack Klapper, MD, Principal Investigator; Stephen H Schechter, MD, Principal Investigator; Olga Klepitskaya, MD, Principal Investigator; Steven Cohen, MD, Principal Investigator; Robert A Hauser, MD, Principal Investigator
Locations (6):
- United States (6):
  - University of Colorado Health Sciences Center, Aurora, Colorado
  - Mile High Research Center, Denver, Colorado
  - CNI Movement Disorders Center, Englewood, Colorado
  - Suncoast Neuroscience Associates, Saint Petersbury, Florida
  - University of South Florida, Tampa, Florida
  - Detroit Clinical Research Center, Novi, Michigan